CLINICAL TRIAL: NCT01924754
Title: GINI: Gardasil Immunogenicity With Needle-free Injection-Safety and Immunogenicity of Gardasil Using IM and ID Needle-free Injection Delivery
Brief Title: Gardasil Immunogenicity With Needle-Free Injection
Acronym: GINI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13366
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-08

CONDITIONS: HPV Seroconversion
Keywords: HPV; Gardasil; seroconversion
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Standard intramuscular injection (NS-IM): HPV vaccination regimen: Standard 3 dose (0.5mL) delivered by standard intramuscular (IM) injection using a needle and syringe (NS-IM)
- PharmaJet needle-free Stratis device (JI-IM): HPV vaccination regimen: Standard 3 dose (0.5mL) delivered by IM injection using the PharmaJet needle-free Stratis device (JI-IM)
- PharmaJet needle-free Tropis device (JI-ID): HPV vaccination regimen: Reduced-dose (0.1 mL) delivered by intradermal injection using the PharmaJet needle-free Tropis device (JI-ID)

SUMMARY:
Using biospecimens collected in a trial by the Thai Red Cross AIDS Research Center that studied two new human papillomavirus (HPV) vaccine delivery regimens, the investigators at UCSF will be testing the serum for antibodies to measure the strength of their response to the vaccine.

DETAILED DESCRIPTION:
Primary Objectives

1. Compared rates of seroconversion and geometric mean titers (GMTs) generated following a 3-dose series of vaccine in women given low doses of vaccine by the intradermal (ID) route with the needle-free injector (NFI) (Group III) to those women given standard doses by the intramuscular (IM) route with a needle and syringe (Group I) at 1 month, 6 months and 12 months following completion of the vaccination series.
2. Compared rates of seroconversion and GMTs generated following a 3-dose series of vaccine in women given standard doses of vaccine by the IM route with the NFI (Group II) to those women given standard doses by the IM route with a needle and syringe (Group I) at 1 month, 6 months and 12 months following completion of the vaccination series.

Serum samples were collected on 4 successive occasions: (1) day zero, prior to the first immunization, (2) at visit 4, one month following the third and final immunization, (3) at visit 5 (12 months) and (4) and at visit 6 (24 months after enrollment). Samples were split, stored and transferred in batch for analysis.

Merck received samples for processing and determined the geometric mean titer of antibodies specific to HPV (types 6, 11, 16, and 18) and results were transferred to the principal investigator. The University of California, San Francisco (UCSF) used a portion of the collected blood samples for pseudovirion-based neutralisation assay (PBNA) analysis conducted at UCSF.

ELIGIBILITY:
Inclusion Criteria:

* Thai women age 18-26 years
* No more than 5 lifetime sexual partners
* HIV-uninfected
* No history of HPV vaccination
* Judged able to complete all of the protocol visits
* No contraindications to vaccination with Gardasil

Exclusion Criteria:

- Does not satisfy all of the inclusion criteria

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study was for women and focused on the safety and immunogenicity of the HPV vaccine. Separate studies will be done in men if the dosing regimens in Groups II or III are shown to be non-inferior to the standard regimen
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- University of California, San Francisco, San Francisco, California, United States
- Thai Red Cross AIDS Research Centre, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 161 women visiting the Thai Red Cross Anonymous Clinic between February 2014 and April 2014 were invited to participate in the study and were screened after providing informed consent. Eleven women were determined to be ineligible
Groups:
- Standard Intramuscular Injection (NS-IM): Human papillomavirus (HPV) vaccination regimen: Standard 3 dose (0.5mL) delivered by standard intramuscular (IM) injection using a needle and syringe
- PharmaJet Needle-free Stratis Device (JI-IM): HPV vaccination regimen: Standard 3 dose (0.5mL) delivered by IM injection using the PharmaJet needle-free Stratis device
- PharmaJet Needle-free Tropis Device (JI-ID): HPV vaccination regimen: Reduced-dose (0.1 mL) delivered by intradermal injection using the PharmaJet needle-free Tropis device
Period: Overall Study
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Started | 50 | 50 | 50
Completed | 49 | 47 | 47
Not Completed | 1 | 3 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Pregnancy | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard Intramuscular Injection (NS-IM): HPV vaccination regimen: Standard 3 dose (0.5mL) delivered by standard intramuscular (IM) injection using a needle and syringe
- Total: Total of all reporting groups
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID) | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23.3 [22.0 to 24.4] | 23.4 [21.2 to 24.9] | 24.5 [22.9 to 25.3] | 23.7 [22.1 to 24.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 50 | 150
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 50 | 50 | 50 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 50 | 50 | 50 | 50
Positive cervical HPV DNA at Baseline [Count of Participants; unit: Participants] — A larger proportion of cases of cervical cancer are caused by infection with HPV types 16 or 18 . HPV types 6 and 11 are low-risk types and cause a majority of anogenital warts in women and men
  Participants
    HPV-6 | 5 | 2 | 1 | 8
    HPV-11 | 0 | 0 | 0 | 0
    HPV-16 | 12 | 5 | 1 | 18
    HPV-18 | 3 | 1 | 3 | 7
Number of HPV genotypes detected at Baseline [Count of Participants; unit: Participants] — Persons can be infected with more than one HPV genotype
  Participants
    1 type | 18 | 4 | 5 | 27
    2 types | 0 | 1 | 2 | 3
    >= 3 types | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Geometric Mean Antibody Concentrations by HPV Type
Description: Geometric mean antibody concentrations above the lower limit of assay detection at baseline were assessed by HPV type
Time Frame: Baseline, up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 50 | 50 | 50
Participants
  HPV-6 | 15 | 12 | 8
  HPV-11 | 4 | 2 | 6
  HPV-16 | 14 | 9 | 8
  HPV-18 | 6 | 4 | 4

2. Primary Outcome: Percentage of Participants With a Demonstrated Seroconversion for HPV 6
Description: The percentage of participants with demonstrated seroconversion generated following a 3-dose series of vaccine for antibodies to HPV 6 at month 7 for the per-protocol efficacy population. The per-protocol efficacy population is defined as as those with month 7 result available, geometric mean antibody concentration below the cutoff level for positivity and undetectable baseline cervical HPV DNA.
Time Frame: Up to 7 months
Measure: Number; unit: percentage of participants
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 32 | 36 | 38
percentage of participants | 100 | 97.2 | 100

3. Primary Outcome: Percentage of Participants With a Demonstrated Seroconversion for HPV 11
Description: The percentage of participants with demonstrated seroconversion generated following a 3-dose series of vaccine for antibodies to HPV 11 at month 7 for the per-protocol efficacy population. The per-protocol efficacy population is defined as as those with month 7 result available, geometric mean antibody concentration below the cutoff level for positivity and undetectable baseline cervical HPV DNA.
Time Frame: Up to 7 months
Measure: Number; unit: percentage of participants
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 45 | 45 | 43
percentage of participants | 100 | 100 | 100

4. Primary Outcome: Percentage of Participants With a Demonstrated Seroconversion for HPV 16
Description: The percentage of participants with demonstrated seroconversion generated following a 3-dose series of vaccine for antibodies to HPV 16 at month 7 for the per-protocol efficacy population. The per-protocol efficacy population is defined as as those with month 7 result available, geometric mean antibody concentration below the cutoff level for positivity and undetectable baseline cervical HPV DNA.
Time Frame: Up to 7 months
Measure: Number; unit: percentage of participants
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 31 | 39 | 39
percentage of participants | 100 | 97.4 | 100

5. Primary Outcome: Percentage of Participants With a Demonstrated Seroconversion for HPV 18
Description: The percentage of participants with demonstrated seroconversion generated following a 3-dose series of vaccine for antibodies to HPV 18 at month 7 for the per-protocol efficacy population. The per-protocol efficacy population is defined as as those with month 7 result available, geometric mean antibody concentration below the cutoff level for positivity and undetectable baseline cervical HPV DNA.
Time Frame: Up to 7 months
Measure: Number; unit: percentage of participants
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 42 | 42 | 42
percentage of participants | 100 | 97.6 | 97.6

6. Primary Outcome: Median Concentration for HPV 6 Over Time
Description: The median (mMU/mL) for HPV 6 at month 7 for the intent to treat population was calculated
Time Frame: Up to 7 months
Measure: Median (Inter-Quartile Range); unit: mMU/mL
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 50 | 50 | 50
mMU/mL
  Baseline | 11 [11 to 15] | 11 [11 to 11] | 11 [11 to 11]
  Month 7 | 449.5 [271 to 750] | 311 [247 to 665] | 259.5 [146 to 395]

7. Primary Outcome: Median Concentration for HPV 11 Over Time
Description: The median concentration (mMU/mL) for HPV 11 at month 7 for the intent to treat population was calculated
Time Frame: Up to 7 months
Measure: Median (Inter-Quartile Range); unit: mMU/mL
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 50 | 50 | 50
mMU/mL
  Baseline | 8 [8 to 8] | 8 [8 to 8] | 8 [8 to 8]
  Month 7 | 517.5 [334 to 769] | 484 [249 to 772] | 387 [197 to 518]

8. Primary Outcome: Median Concentration for HPV 16 Over Time
Description: The median concentration (mMU/mL) for HPV 16 at month 7 for the intent to treat population was calculated
Time Frame: Up to 7 months
Measure: Median (Inter-Quartile Range); unit: mMU/mL
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 50 | 50 | 50
mMU/mL
  Baseline | 11 [11 to 26] | 11 [11 to 11] | 11 [11 to 11]
  Month 7 | 2243.5 [1669 to 4227] | 2054.5 [1297 to 3332] | 1482 [730 to 2584]

9. Primary Outcome: Median Concentration for HPV 18 Over Time
Description: The median concentration (mMU/mL) for HPV 18 at month 7 for the intent to treat population was calculated
Time Frame: Up to 7 months
Measure: Median (Inter-Quartile Range); unit: mMU/mL
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 50 | 50 | 50
mMU/mL
  Baseline | 10 [10 to 10] | 10 [10 to 10] | 10 [10 to 10]
  Month 7 | 412.5 [193 to 768] | 414.5 [166 to 610] | 372.5 [142 to 578]

10. Primary Outcome: Geometric Mean Concentration Ratio of NS-IM Versus the PharmaJet Groups by HPV Type
Description: The Geometric Mean Concentration Ratio (GMCR) and 95% confidence interval for both NS-IM versus JI-IM and NS-IM versus JI-ID was computed for the intent to treat population. Non-inferiority for arms JI-IM and JI-ID was defined as geometric mean concentration ratio (GMCR) <1.5 of NS-IM at month 7
Time Frame: Up to 7 months
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
Number analyzed (Participants) | 50 | 50
ratio
  HPV-6 | 1.37 [0.90 to 2.08] | 1.84 [1.30 to 2.61]
  HPV-11 | 1.36 [0.94 to 1.96] | 1.61 [1.19 to 2.17]
  HPV-16 | 1.47 [0.97 to 2.24] | 1.97 [1.34 to 2.90]
  HPV-18 | 1.23 [0.79 to 1.91] | 1.52 [0.99 to 2.33]

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Immediate complaints (noted within 30 minutes after vaccination), solicited adverse events (local and systemic) from the first day after vaccination until 7 days after the vaccination as reported on diary cards, and unsolicited reported adverse events during the study
Arm/Group | Standard Intramuscular Injection (NS-IM) | PharmaJet Needle-free Stratis Device (JI-IM) | PharmaJet Needle-free Tropis Device (JI-ID)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50 | 3/50 | 2/50
Other Adverse Events (participants affected / at risk) | 45/50 | 46/50 | 36/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Intramuscular Injection (NS-IM) (N=50) | PharmaJet Needle-free Stratis Device (JI-IM) (N=50) | PharmaJet Needle-free Tropis Device (JI-ID) (N=50)
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Intramuscular Injection (NS-IM) (N=50) | PharmaJet Needle-free Stratis Device (JI-IM) (N=50) | PharmaJet Needle-free Tropis Device (JI-ID) (N=50)
Injection site pain (Investigations) | 44 | 44 | 23
Swelling (Investigations) | 21 | 32 | 21
Arm movement limitation (Musculoskeletal and connective tissue disorders) | 35 | 33 | 9
Erythema (Investigations) | 14 | 23 | 27
Itching (Skin and subcutaneous tissue disorders) | 6 | 14 | 15
Induration (Investigations) | 7 | 20 | 27
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 9 | 7
Headache (Nervous system disorders) | 15 | 11 | 4
Chills (General disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 12 | 14 | 6
Fatigue (General disorders) | 26 | 20 | 9
Nausea (Gastrointestinal disorders) | 6 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 31 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No